CLINICAL TRIAL: NCT05929287
Title: A Comparison Between Personalized and Adaptive Tablet-based Cognitive Training and Paper-and-pencil Cognitive Training: a Randomized Controlled Trial With Community Dwelling Stroke Patients
Brief Title: Comparing Personalized and Adaptive Cognitive Training Methods Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Responsible Party: Principal Investigator, Sergi Bermúdez i Badia, Associate Professor at the University of Madeira and Senior Researcher at NOVA LINCS, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43/2019
Record Dates: First submitted 2023-06-05; First posted 2023-07-03 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Cognitive Training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants won't be aware of which group they are randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1. Tablet-based CT (NeuroAIreh@b) (Experimental): Participants in the NeuroAIreh@b group will perform tablet-based CT tasks personalized to their underlying deficits and performance in each iteration.
  Biweekly 30-minute sessions until reaching 12 sessions.
  Interventions: Procedure: Tablet-based CT
- Experimental group 2. Paper-and-pencil CT (Task Generator). (Experimental): Participants in the paper and pencil group will perform CT tasks personalized to their cognitive deficits (according to the MoCA) and generated automatically through the Task Generator website (https://neurorehablab.arditi.pt/TaskGenerator/).
  Biweekly 30-minute sessions until reaching 12 sessions.
  Interventions: Procedure: Paper-and-pencil CT group
- passive control group (Waiting-list). (No Intervention): Participants in this group will not be enrolled in any intervention during the course of the study. At the end of the study, participants can integrate a CT intervention of their choice (e.g., CT through the NeuroAIreh@b platform or the TG).

INTERVENTIONS:
Procedure: Tablet-based CT — This group will perform digital CT tasks.
  Arms: Experimental group 1. Tablet-based CT (NeuroAIreh@b)
Procedure: Paper-and-pencil CT group — This group will perform paper-and-pencil CT tasks.
  Arms: Experimental group 2. Paper-and-pencil CT (Task Generator).

SUMMARY:
This study aims to assess the efficacy of two cognitive training programs - one tablet-based (NeuroAIreh@b) and one in paper-and-pencil format (Task Generator) - in improving cognitive and noncognitive outcomes among community-dwelling stroke survivors.

This study will include a waiting-list control group to assess the impact of these interventions and provide further insights into their potential for stroke survivors.

DETAILED DESCRIPTION:
The investigators plan to conduct a multicentric clinical trial with 45 participants randomly assigned to one of three groups. The study will have three arms, with each group receiving one of the following interventions: table-based cognitive training (NeuroAIreh@b), paper-and-pencil cognitive training (Task Generator) or no intervention (waiting-list control group). The latter group will not receive intervention during the study but will be offered the opportunity to participate in one of the cognitive training programs after completing the study. Additionally, the investigators will assess participants at three different time points: before the intervention (pre-intervention), immediately after the intervention (post-intervention), and three months after the intervention (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis;
* Maximum age: 75 years old;
* Education: at least three years of formal education;
* Relatively preserved language abilities (expressive and receptive language);
* Residing in the community;
* Availability to go to the hospital 2x/week;
* Preserved visual and auditory acuity;
* Physically able to operate the tablet and perform the paper-and-pencil training;
* Motivation to participate.

Exclusion Criteria:

* Diagnosis of concomitant neurological and/or psychiatric disorders;
* Hemianopsia;
* Unilateral neglect;
* Aphasia syndromes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months).
  change from baseline to post-intervention, and baseline to follow-up, in the MoCA; Min score=0; Max score=30; Higher are indicative of a better performance;
Symbol Search and Digit Symbol (WAIS-III) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months)
  change from baseline to post-intervention, and baseline to follow-up, in both the Symbol Search and the Digit Symbol (WAIS-III); Min score=0; Max score=Dependent on participants' performance during the 120 seconds tasks. Higher scores in both subtests are indicative of a better performance.
Toulouse-Piéron Cancellation Test (TP) | : baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months)
  change from baseline to post-intervention, and baseline to follow-up, in the TP; Min and Max scores=dependent on participants' performance during 10 minutes. A higher work efficiency index is indicative of a better performance, while a higher dispersion index is indicative of a worse performance.
Rey-Complex Figure Test (ROCFT) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months)
  Change from baseline to post-intervention, and baseline to follow-up, in the ROCFT; Min score=0; Max score=36. Higher scores on both the copy trial and 3-minutes immediate recall trial are indicative of a better performance.
Auditory Verbal Learning Test (AVLT) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months)
  Change from baseline to post-intervention, and baseline to follow-up, in the AVLT; Min score=0; Max score=varies across trials (5 immediate recall trials: 75 points; 1 delayed recall trial: 15 points; 1 delayed recognition task: 30 points). Higher scores are indicative of a better performance.
Verbal Fluency Tests | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months).
  Change from baseline to post-intervention, and baseline to follow-up, in the verbal fluency tests; Min score=0; Max score=dependent on participants' performance during the 1-minute task. Higher scores on the verbal fluency tests are indicative of a better performance.

SECONDARY OUTCOMES:
Subjective Memory Complaints Questionnaire (SMCQ) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months).
  Change from baseline to post-intervention, and baseline to follow-up, in the SMCQ; Min score=0; Max score=21; Higher scores are indicative of worse self-perceived memory decline.
Hospital Anxiety and Depression Scale (HADS) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months).
  Change from baseline to post-intervention, and baseline to follow-up, in the HADS; Min score=0; Max score=42; Higher scores are indicative of worse self-perceived emotional stability.
Quality of Life after Brain Injury (QOLIBRI) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months)
  Change from baseline to post-intervention, and baseline to follow-up, in the QOLIBRI; Min score=0; Max score=100; Higher scores are indicative of greater self-perceived quality of life.
Adults and Older Adults Functional Assessment Inventory (IAFAI) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months).
  Change from baseline to post-intervention, and baseline to follow-up, in the IAFAI; Min=0; Max=100; Higher scores are indicative of a worse self-reported functional disability.
Motivation for Traumatic Brain Injury Rehabilitation Questionnaire (MOT-Q) | baseline (1 week before the beginning of the intervention), post-intervention (7 weeks), and follow-up (1-month and 3-months).
  Change from baseline to post-intervention, and baseline to follow-up, in the MOT-Q; Min=-62; Max=62; Higher scores indicate higher motivation for rehabilitation.

CONTACTS AND LOCATIONS:
Locations (1):
- ARDITI, Edif. Madeira Tecnopolo, Caminho da Penteada piso 2, 9020-105 Funchal, Funchal, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camara J, de Aguiar SC, Paulino T, Faria AL, Bermudez I Badia S, Vilar M, Ferme E. Comparing adaptive tablet-based cognitive training and paper-and-pencil cognitive training: a pilot randomized controlled trial with community-dwelling stroke survivors. Int J Clin Health Psychol. 2025 Jul-Sep;25(3):100627. doi: 10.1016/j.ijchp.2025.100627. Epub 2025 Sep 25. PMID 41070261

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT05929287/Prot_ICF_000.pdf